CLINICAL TRIAL: NCT03058120
Title: Henry Ford Heart Score Randomized Trial: Rapid Discharge of Patients Evaluated for Possible Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Tiberio Frisoli, MD, Member of Heart and Vascular Institute in the Division of Cardiology, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB 8558
Record Dates: First submitted 2017-02-14; First posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Chest Pain; Heart Attack; Coronary Artery Disease
MeSH Terms: conditions — Chest Pain; Myocardial Infarction; Coronary Artery Disease | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress testing (No Intervention): Patient with chest pain, low risk by modified HEART score, undergoes whatever admission and stress testing plan is determined by ED and inheriting decision unit physicians.
- Early discharge (Active Comparator): Patient with chest pain, low risk by modified HEART score, is discharged from the emergency room without admission nor stress testing.
  Interventions: Other: Deferral of admission for stress test

INTERVENTIONS:
Other: Deferral of admission for stress test — Early discharge; admission and stress test are deferred.
  Arms: Early discharge

SUMMARY:
This was a prospective randomized, controlled trial designed to quantify the reduction in cost and length of stay of early discharge of emergency department patients evaluated for acute myocardial infarction, who are deemed to be low risk based on a modified HEART score (a score that incorporates troponin biomarker, ecg, patient characteristics, and physician clinical judgment).

DETAILED DESCRIPTION:
This was a prospective randomized, controlled trial conducted from February 2014 to May 2015 designed to quantify the reduction in cost and length of stay of early discharge of emergency department patients evaluated for acute myocardial infarction, in those deemed to be low risk based on a modified HEART score. Our study enrolled only those deemed low risk, as these are the patients we believe best served by utilization of the HEART score decision aid.

A total of 105 patients evaluated for AMI in the ED with a modified HEART score ≤ 3 (which includes cardiac troponin I < 0.04 ng/ml at 0 and 3 hours) were randomized to immediate discharge (n = 53) vs management in an observation unit with stress testing (n = 52).

The primary endpoints were 30-day total cost and length of stay. Secondary endpoints were all-cause death, nonfatal AMI, rehospitalization for evaluation of possible AMI, and coronary revascularization at 30 days.

That such an early discharge strategy would decrease cost and length of stay is intuitively expected; our goal was to quantify such a reduction.

ELIGIBILITY:
Inclusion Criteria:

* patients 21 years or older
* patients who presented to the Emergency Department with symptoms suspicious for AMI.
* patients for whom the ED physician's intention to send the patient to the observation unit for stress testing

Exclusion Criteria:

* Cardiac Troponin I > 0.04 ng/mL at 0 or 3 hours
* clinical presentation warranting admission
* inability or unwillingness to consent
* trauma as etiology of presenting symptoms.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-02-19 (Actual); Primary Completion 2015-05-08 (Actual); Study Completion 2015-05-08 (Actual)

PRIMARY OUTCOMES:
Cost of hospitalization | 30 days
  Total charges accrued during index hospitalization, as well as costs related to index hospitalization up to 30 days after index discharge
Length of stay | up to 1 week
  Total length of stay of index hospitalization

SECONDARY OUTCOMES:
30-day MACE | 30 days after index hospitalization
  Death, non-fatal myocardial infarction, stroke

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frisoli TM, Nowak R, Evans KL, Harrison M, Alani M, Varghese S, Rahman M, Noll S, Flannery KR, Michaels A, Tabaku M, Jacobsen G, McCord J. Henry Ford HEART Score Randomized Trial: Rapid Discharge of Patients Evaluated for Possible Myocardial Infarction. Circ Cardiovasc Qual Outcomes. 2017 Oct;10(10):e003617. doi: 10.1161/CIRCOUTCOMES.117.003617. PMID 28954802